CLINICAL TRIAL: NCT04299061
Title: The Effect of the Physical Activity and Healthy Living Elective Courses on Physical Activity Level and Awareness Among University Students Educating in Different Departments
Brief Title: Effect of the Physical Activity Courses on the Physical Activity Level at University Students
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic, sufficient number of participants could not be received.
Sponsor: Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Gamze Ertürk, PhD Student, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FASYD-1
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity Level; Physical Activity Awareness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Diagnostic Test: International Physical Activity Questionnaire; Diagnostic Test: Pittsburgh Sleep Quality Index; Other: Physical Activity Awareness Questionnaire - prepared by the researchers; Diagnostic Test: Perceived Stress Scale

INTERVENTIONS:
Diagnostic Test: International Physical Activity Questionnaire — This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. Walking = 3.3 METs Moderate Intensity = 4.0 METs Vigorous Intensity = 8.0 METs Total MET-minutes/week = Walk (METs*min*days) + Mod (METs*min*days) + Vig (METs*min*days)
  1. Low: • No activity is reported OR • Some activity is reported but not enough to meet Categories 2 or 3. 2. Moderate: • 3 or more days of vigorous activity of at least 20 minutes per day OR • 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR • 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-minutes/week. 3. High: • Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week
Diagnostic Test: Pittsburgh Sleep Quality Index — The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month.The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5"or greater indicates a "poor" sleeper.
Other: Physical Activity Awareness Questionnaire - prepared by the researchers — It consists of 13 questions to assess the physical activity level awareness of students. The questionnaire was prepared by the researchers therefore it does not have a validation.
Diagnostic Test: Perceived Stress Scale — The Perceived Stress Scale (PSS) is a classic stress assessment instrument that helps understand how different situations affect feelings and perceived stress. The questions in this scale ask about feelings and thoughts during the last month. It consists of 14 questions.

SUMMARY:
The aim of our study is to evaluate the level of physical activity and awareness of physical activity among university students studying in a department other than health sciences and who have taken courses on "physical activity, exercise, healthy life".

According to the results of the study, the perceptions of students from different departments on physical activity and exercise will be compared and the effects of the courses they have taken on students' attitudes of daily physical activity will be examined.

Our hypothesizes are:

1 . A course such as an exercise, physical activity or wellness increases the awareness and physical activity level of students studying in different branches.

2. Stress and sleep problems are less common among students who do regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Being a student in departments of lawyer, engineering and architecture in university
* Participation in courses is compulsory
* For the study group; having taken physical activity, exercise, wellness classes as compulsory or optional in their university
* For the control group; not taking physical activity, exercise, wellness lessons in their university

Exclusion Criteria:

* Being a student in other departments

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | Baseline of the study
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. Walking = 3.3 METs Moderate Intensity = 4.0 METs Vigorous Intensity = 8.0 METs Total MET-minutes/week = Walk (METs*min*days) + Mod (METs*min*days) + Vig (METs*min*days). 1. Low: • No activity is reported OR • Some activity is reported but not enough to meet Categories 2 or 3. 2. Moderate: • 3 or more days of vigorous activity of at least 20 minutes per day OR • 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR • 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-minutes/week. 3. High: • Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week
Physical Activity Awareness Questionnaire - prepared by the researcher | Baseline of the study
  It consists of 13 questions to assess the physical activity level awareness of students. The questionnaire was prepared by the researchers so it does not have a validation. Questions are about determined the difference between meanings of exercise and physical activity. For example:
  Mark it as yes, no or not know.
  1. Physical activity and exercise mean the same thing.
  2. Physical activity is a subcategory of exercise.
Pittsburgh Sleep Quality Index | Baseline of the study
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Perceived Stress Scale | Baseline of the study
  The Perceived Stress Scale (PSS) is a 14-item self-report measure designed to assess "the degree to which situations in one's life are appraised as stressful. Each item is rated on a 5-point scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often) and summed to create a total score. PSS-14 has strong internal consistency (α = .84 to .86) and good test-retest reliability (r = .85 over a 2-day period, r = .55 over a 6-week period.

IPD SHARING:
Plan to Share IPD: Undecided